CLINICAL TRIAL: NCT01372670
Title: Hydroxyzine Effects on Meal-Related Anxiety in Underweight Adolescents and Young Adults Diagnosed With an Eating Disorder - A Pilot Study
Brief Title: Does Hydroxyzine Decrease Anxiety in Underweight Patients Diagnosed With an Eating Disorder
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Why Stopped: Due to unforseen recruiting difficulties, the study was closed.
Sponsor: HealthPartners Institute (Other)
Collaborators: Park Nicollet Eating Disorder Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Triple | Purpose: Treatment
Other Study IDs: 04091-11
Record Dates: First submitted 2011-06-10; First posted 2011-06-14 (Estimated); Last update posted 2016-11-15 (Estimated); Status verified 2016-02

CONDITIONS: Anxiety in Those Patients With Anorexia Nervosa; Eating Disorder Not Otherwise Specified, BMI (<=18)
Keywords: Treating meal related anxiety
MeSH Terms: interventions — Hydroxyzine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Hydroxyzine (Experimental): Hydroxyzine given TID
  Interventions: Drug: Hydroxyzine; Drug: hydroxyzine HCL
- Sugar Pill (Placebo Comparator): Placebo given 3 times per day
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Hydroxyzine — Study medications (hydroxyzine/placebo) will be dosed based on participant's weight. Dosing will be according to the following body weight ranges:
  15-29 Kg 10 mg TID 30-44 Kg 20 mg TID
  ≥ 45 Kg 30 mg TID
  Arms: Hydroxyzine
Drug: hydroxyzine HCL — hydroxyzine HCL dosed on weight given 3x per day
  Arms: Hydroxyzine
Other: Placebo — Placebo given 3 times per day
  Arms: Sugar Pill

SUMMARY:
The purpose of this study is to determine the effectiveness of hydroxyzine in the treatment of meal-related anxiety in adolescents and young adults 8 to 25 years of age diagnosed with an eating disorder who are underweight. The investigators want to find out if hydroxyzine given before meals will improve meal-related anxiety compared to no hydroxyzine.

DETAILED DESCRIPTION:
This study is a practiced-based pilot study in follow-up to clinical observations made by our treatment team that hydroxyzine attenuates meal-related anxiety and improves treatment adherence in patients with a diagnosis of Anorexia Nervosa (AN) (excluding the amenorrhea criterion) or Eating Disorder Not Otherwise Specified (EDNOS) specifically with low BMI (≤ 18). To our knowledge, hydroxyzine has never been formally investigated in treating meal-related anxiety and improving outcomes in patients with AN or EDNOS specifically with low BMI (≤ 18).

ELIGIBILITY:
Inclusion Criteria:

* Admitted to the Intensive Structured Living Unit (ISL) at Melrose Institute for treatment of an eating disorder that meets DSM-IV criteria for Anorexia Nervosa (excluding the amenorrhea criterion), or Eating Disorder Not Otherwise Specified, specifically with BMI (≤ 18)
* Age 8-25 years old at admission to ISL.
* Weight ≥ 15 kg at admission to ISL.
* Stable psychotropic and/or sedative medications for at least (≥) 6 weeks

Exclusion Criteria:

* Age < 8 years
* Age ≥ 25 years
* Weight < 15 kg at admission to ISL
* Prolonged QT interval on ECG at admission to ISL
* Current substance or alcohol abuse or dependence
* Malabsorption syndrome or inability to take oral medications
* History of hydroxyzine intolerance or hypersensitivity
* History of Type 1 Diabetes Mellitus
* History of angle closure glaucoma
* Currently on another clinical trial
* Pregnancy

Ages: 8 Years to 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 0 (Actual)
Dates: Start 2012-01; Primary Completion 2013-04 (Actual); Study Completion 2013-04 (Actual)

PRIMARY OUTCOMES:
Self-reported anxiety | 3 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Marcus Westerman, MD, PhD, Principal Investigator — Park Nicollet Melrose Institute
Locations (1):
- Melrose Institute, Minneapolis, Minnesota, United States